CLINICAL TRIAL: NCT04071444
Title: Exploring the Predictors of Constipation and the Effects of a Baduanjin Program on the Symptoms of Constipation in Adults With Chronic Schizophrenia
Brief Title: Exploring the Effects of a Baduanjin Program on the Symptoms of Constipation in Patients With Schizophrenia Spectrum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Tri-Service General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2-107-05-114
Record Dates: First submitted 2019-08-25; First posted 2019-08-28 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2018-03

CONDITIONS: Randomized Controlled Trial
Keywords: Baduanjin program; constipation; intestinal peristalsis; schizophrenia spectrum
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Intervention Model Description: The participants were divided into experimental and control groups through block randomization.
Who Masked: Participant
Masking Description: The data of Intestinal Peristalsis in four quadrants were collected by a research assistant.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baduanjin program (Experimental): The entire program continued for 6 months (December, 2018 to July, 2019), and the intervention was performed for 60 min 3 times per week; particular attention was paid to the disease characteristics of the patients with chronic schizophrenia and to preventing excessive fatigue. Every session began with a 20-min warm-up, followed by 20 min of Baduanjin program, and ended with a cool-down session. The participants were instructed, with the assistance of a video, to practice Baduanjin program in a group by two authors who are experienced in the psychiatric nurses and had been trained in this program.
  Interventions: Other: Baduanjin program
- Control group (No Intervention): The control group (CG) received routine care.

INTERVENTIONS:
Other: Baduanjin program — The entire program continued for 6 months (December, 2018 to July, 2019), and the intervention was performed for 60 min 3 times per week; particular attention was paid to the disease characteristics of the patients with chronic schizophrenia and to preventing excessive fatigue. Every session began with a 20-min warm-up, followed by 20 min of Baduanjin program, and ended with a cool-down session. The participants were instructed, with the assistance of a video, to practice Baduanjin program in a group by two authors who are experienced in the psychiatric nurses and had been trained in this program.
  Arms: Baduanjin program

SUMMARY:
Patients with schizophrenia spectrum have been suffering from constipation due to long-term use of psychotropic medications and changes in physical activity and eating habits caused by diseases.

Aim this study was to examine the effectiveness of Baduanjin program in improving the symptoms of intestinal peristalsis and constipation in patients with psychosis.

Method:A randomized controlled trial was conducted in tow psychiatric centers in northern Taiwan.The experimental group was provided with an 8- session Baduanjin program for 24 weeks (1 hour, thrice times per week), while the control group received routine care.

DETAILED DESCRIPTION:
This study was conducted in two psychiatric center. Residents in one of psychiatric center were allowed to walk for 20 min after dinner every day, and each unit residents rare active. In this study, patients on the schizophrenia spectrum were invited to receive screening for constipation syndrome. A total of 275 patients agreed to undergo the screening. In total of 112 patients satisfied the inclusion criteria, and 58 patients consented to participate in the experiment.

Each participant was assigned one number from 1 to 112 by the first author. The second author enrolled participants. They were randomized to either Baduanjin program group or routine care group in a 1:1 ratio using blocked randomization having a block size of 3. Patients in the experimental group (EG) participated in the Baduanjin intervention in a privacy setting", which involved 60-min sessions 3 times per week, 1 hour after dinner between 6 and 7 pm; the entire program continued for 24 weeks. The control group (CG) received routine care. The outcome indicators for this intervention program involved the risk factors for constipation, constipation symptoms, and Intestinal Peristalsis.

ELIGIBILITY:
Inclusion Criteria:

* Comply with the diagnosis of the spectrum.
* Have the willingness to participate in the study and could read, communicate and cooperate with the completion of the consent form and questionnaire.
* The age is 20 to 64 years old.
* No need for any assistance in walking, and the gait is stable.
* Appeared more than 2 times in the past month for more than 3 consecutive days without resolving or routine use of laxatives

Exclusion Criteria:

* Diagnosis is organic brain disease, alcohol and substance abuse.
* There have been problems with gastrointestinal bleeding or lesions.
* Have a history of extensive abdominal surgery or gastrointestinal surgery.
* There are medical considerations and medical expenses reduction activities.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2018-10-08 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Changes in Intestinal Peristalsis | 3 months and 6 months
  Change from Baseline bowel movement of four quadrants of abdomen at 3 months and 6 months

SECONDARY OUTCOMES:
Changes in Constipation Assessment Scale | 3 months and 6 months
  Change from Baseline Constipation Assessment Scale at 3 months and 6 months. The nine symptoms evaluated included: bloating, increased gas delivery in the rectum, decreased / increase frequency of bowel movements, oozing water, rectal obstruction or pressure, bowel movements combined with rectal pain, low bowel movements, and inability to defecate. 3 points scoring method (0-2), 0 is no problem, 1 is a bit problem, 2 is a serious problem. The maximum total score is 18.
Change in Patient Assessment of Constipation Symptoms | 3 months and 6 months
  Change from Baseline Patient Assessment of Constipation Symptoms at 3 months and 6 months. The 12 items are divided into 3 subscales: 4 items for abdominal symptoms, 3 items for rectal symptoms, and 5 items for fecal symptoms. Patient Assessment of Constipation Symptoms Scale items are rated on a 5-point scale ranging from 0 to 4 based on severity of each item. The maximum total score is 48.

CONTACTS AND LOCATIONS:
Overall Officials: Chiu-Yueh Yang, PhD, Principal Investigator — Yang Ming National University; Li-Ru Wang, MSN, Study Director — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan